CLINICAL TRIAL: NCT03019614
Title: An Open Label, Randomised, Single Dose, 3-period Crossover Study in Healthy Volunteers to: a) Compare the Pharmacokinetics of Chronocort® Formulations Versus Immediate Release Hydrocortisone, and (b) Determine the Dose Proportionality of Chronocort® Formulations
Brief Title: An Open Label Study in Healthy Volunteers to Compare Chronocort® to Hydrocortisone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DIUR-001
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Adrenal Hyperplasia; Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Adrenal Insufficiency | interventions — Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Volunteers in group 1 received the following interventions:
  Chronocort® 30 mg given at night (~ 23:00h) as a combination of one 10mg capsule and one 20mg capsule (n=18).
  Chronocort® 30mg given as one 20mg capsule at night (~ 23:00h) and as one 10mg capsule in the morning (~ 7:00h) following the initial night-time dose (n=18).
  Hydrocortisone 30mg given at night (~ 23:00h) given as three 10mg tablets (n=18).
  Each administration of IMP was separated by a washout period of at least 7 days.
  Interventions: Drug: Hydrocortisone; Drug: Chronocort
- Group 2 (Experimental): Volunteers in group 2 received the following interventions:
  Chronocort® 5mg given at night (~ 23:00h) as one 5mg capsule (n=12).
  Chronocort® 10mg given at night (~ 23:00h) as one 10mg capsule (n=12).
  Chronocort® 20mg given at night (~ 23:00h) as one 20mg capsule (n=12).
  Each administration of IMP was separated by a washout period of at least 7 days.
  Interventions: Drug: Chronocort

INTERVENTIONS:
Drug: Hydrocortisone — Generic hydrocortisone
  Arms: Group 1
Drug: Chronocort — Modified formulation of hydrocortisone

SUMMARY:
This was an open label, randomized, single dose, three period crossover pharmacokinetic study of Chronocort® in 30 healthy male volunteers. The study was conducted in smaller sub groups (Group 1, n=18 and Group 2, n=12).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between 18 and 60 years of age, inclusive (at screening).
* Subjects with a Body Mass Index (BMI) of 21-28. Body Mass Index = Body weight (kg) / (Height (m))2.
* Subjects with no clinically significant abnormal serum biochemistry, haematology and urine examination values within 14 days of the start of the study. The parameters measured included those shown in Appendix 3 of the Study Protocol.
* Subjects with a negative urinary drugs of abuse screen (including alcohol), determined within 14 days of the start of the study.
* Subjects with negative HIV and Hepatitis B and C results.
* Subjects with no clinically significant abnormalities in 12-lead electrocardiogram (ECG) determined within 14 days of the start of the study.
* Subjects with no clinically-significant deviation outside the normal ranges for blood pressure and pulse measurements.
* Subjects and sexual partners must have used effective contraception methods during the trial and for 3 months after the last dose, for example:

  * Oral contraceptive + condom
  * Intra-uterine device (IUD) + condom
  * Diaphragm with spermacide + condom
* Subjects must have been available to complete the study.
* Subjects must have satisfied a medical examiner about their fitness to participate in the study.
* Subjects must have provided written informed consent to participate in the study.

Exclusion Criteria:

* A clinically significant history of gastrointestinal disorder likely to influence drug absorption.
* Receipt of regular medication within 14 days of the first study day (including high dose vitamins, dietary supplements or herbal remedies).
* Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
* A clinically significant history of previous allergy / sensitivity to Hydrocortisone.
* A clinically significant history of drug or alcohol abuse.
* Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
* Participation in a New Chemical Entity clinical study within the previous 16 weeks or a marketed drug clinical study within the previous 12 weeks.
* Subjects who had consumed more than 2 units of alcohol per day within seven (7) days prior to the first dose or had consumed any alcohol within the 48 hour period prior to the first dose.
* Donation of 450ml or more blood within the previous 12 weeks.
* Subjects who worked shifts (i.e. regularly alternated between days, afternoons and nights).

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Derived pharmacokinetic parameter: Tmax | 24 hours
  Tmax measures the time at which Cmax - maximum serum concentration - is observed
Derived pharmacokinetic parameter: Tlag | 24 hours
  Tlag measures the delay between dosing and being able to observe the drug/metabolite within the sampling area (e.g., blood serum)
Derived pharmacokinetic parameter: Cmax | 24 hours
  Cmax measures the time taken for the drug/metabolite to reach maximum serum concentration
Derived pharmacokinetic parameter: AUC(0 - t) (Area under the curve) | 24 hours
  Area under the serum concentration versus time curve from time
Derived pharmacokinetic parameter: AUC(0-∞)(Area under the curve) | 24 hours
  Area under the serum concentration versus time curve from time = 0h extrapolated to infinity
Derived pharmacokinetic parameter: CL | 24 hours
  Time to drug clearance
Derived pharmacokinetic parameter: T1/2 | 24 hours
  Time required to reach 1/2 Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Febbraro, Principal Investigator — Simbec Research

IPD SHARING:
Plan to Share IPD: No